CLINICAL TRIAL: NCT06763614
Title: A Randomised Controlled Study of Dog Assisted Therapy: Comparing a Short and a Long Version Program for Patients with Fetal Alcohol Spectrum Disorder.
Brief Title: Dog Assisted Therapy: Comparing Duration Treatments for Patients with Fetal Alcohol Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Fundacion Probitas (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAT-VH-2023
Record Dates: First submitted 2024-07-22; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2023-07

CONDITIONS: Fetal Alcohol Spectrum Disorders
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- A Randomised Controlled Study Of Dog Assisted Therapy (Experimental): We tested 8 week dog assisted therapy for patients with FASD vs 16 week treatment for patients with FASD
  Interventions: Behavioral: Dog assisted therapy - animal interventions

INTERVENTIONS:
Behavioral: Dog assisted therapy - animal interventions — Animal Assisted Therapy is when animals are used in goal directed treatment sessions. These goals are working emotionalaspects pf childres and adolescents with SAF

SUMMARY:
The objective of the present study was to assess the efficacy of a shorter version program of Dog Assisted Therapy (DAT) (8 sessions) compared to a longer version (16 sessions) for children and adolescents with Fetal Alcohol Syndrome (FASD). We evaluated the impact of DAT on social skills, internalizing and externalizing problems, quality of life, severity of the disorder and emotional well-being of parents. We conducted a randomized controlled trial in a cohort of 55 patients with FASD.

DETAILED DESCRIPTION:
FASD can be classified into three subtypes. FAS is identified by (1) facial abnormalities, (2) growth deficits, abnormal brain development, or irregularities in neurophysiology, and (3) neurobehavioral issues. Partial Fetal Alcohol Spectrum Disorder (FASD) shares similarities but presents with fewer physical characteristics, while Alcohol-Related Neurobehavioral Disorder (ARND) solely exhibits neurobehavioral symptoms without facial anomalies.

Previous research has highlighted the effectiveness of psychological intervention programs focused on emotional regulation for individuals with FASD. Similarly, studies have emphasized the benefits of interventions targeting social skills. These interventions have been shown to result in reductions in externalizing behaviors, with social skills training specifically correlating with improvements in social competence and a decrease in problematic behaviors Recently a new form of behavioral therapy has been gaining popularity in improving the physical and mental health of young adults, known as Animal Assisted Therapy (AAT). Animal Assisted Therapy lays its foundation in human attachment theory and social cognitive theory where it is argued that animals can be potentially viewed as a transitional attachment object and thus aid to improve psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:all participants needed to have stable doses of medication for at least two months before the study and agree not to seek out any other psychiatric or psychological treatment during the study.

-

Exclusion Criteria:Patients who were not behaviorally stable, presented agressive behavior or required more intensive treatment (hospitalization or day hospital) were excluded.

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Wechsler Intelligence Scale for Children | Once- Pre intervention week 1 - Post intervention in week 16
  Intellectual Quotient
Child Behavior Checklist (CBCL by Achenbach) | Once- Pre intervention week 1 - Post intervention in week 16
  Internalizing/ Externalizing Symptoms maximum scores for symptom severity 113
Social Skills Improvement System-Parent Form (SSIS-P) | Once- Pre intervention week 1 - Post intervention in week 16
  Social skills assessment - 0 to 60 max scotring
KidScreen 27- 0 maximum 135 - highest severity symptoms at 135 | Once- Pre intervention week 1 - Post intervention in week 16
  Quality of life assesment
Clinical Global Impression Scale for Severity.0 to 7 (7 most severely ill). | Once- Pre intervention week 1 - Post intervention in week 16
  Severity of FASD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Josep Antoni Ramos Quirogfa, MD-PHD, Study Director — Comitè Ètic d'Investigació Clínica HUVH Barcelona, Barcelona Spain
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The data collected from the patients evaluated in our hospital will be stored in the medical records of Vall d'Hebron University Hospital, as well as in a computerized database that allows for analysis. Rigorous confidentiality of the data will be maintained in accordance with current regulations in Spain (Ley Orgánica de Protección de Datos). To analyze the final data from the three hospitals, each patient will be coded (anonymous code) to facilitate data processing.